CLINICAL TRIAL: NCT04814004
Title: Clinical Study of CAR-iNKT Cells in the Treatment of Relapsed/Refractory/High-risk B-cell Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai Lin Xu; Jun Nian Zheng (Other)
Collaborators: North Jiangsu People's Hospital (Unknown); The First People's Hospital of Changzhou (Other); Nantong University (Other); First Affiliated Hospital of Zhejiang University (Other); Affiliated Hospital of Jiangsu University (Other); Huai 'an First People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Kai Lin Xu; Jun Nian Zheng, Principal Investigator, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2021-KL062
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Acute Lymphoblastic Leukemia; B-cell Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hCD19.IL15.CAR-iNKT cells (Experimental): Dose escalation follows the accelerated titration and the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Drug: hCD19.IL15.CAR-iNKT

INTERVENTIONS:
Drug: hCD19.IL15.CAR-iNKT — Universal hCD19.IL15.CAR-iNKT cells by a single infusion intravenously will be given in escalating doses.

SUMMARY:
This study aims to evaluate the safety and feasibility of hCD19.IL15.CAR-iNKT cells in treating patients with relapsed/refractory/high-risk B-cell tumors.

DETAILED DESCRIPTION:
CD19 CAR-T has been shown to treat a variety of refractory or recurrent B-cell tumors. Because most CAR-T cells are generated from the patient's own T cells and are individualized products, and there are individual differences between patients, the generation of customized CAR-T cells is an expensive and time-consuming process. Universal CAR- iNKT cells are an ideal product for cell therapy. In this study, we prepared universal iNKT cells expressing hCD19 CAR and IL-15 to treat refractory, relapsed, or high-risk B-cell tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 5-70 years;
* The patient's ECOG score was ≤2, and the expected survival time of > was 12 weeks.
* The patient was diagnosed with B-cell tumor by pathological and histological examination and had no effective treatment options, such as recurrence after chemotherapy or hematopoietic stem cell transplantation. Or the patient voluntarily chooses the infusion of CAR-INKT cells as the first treatment.
* B cell tumors include the following three types:

  1. B-cell acute lymphocytic leukemia (B-ALL);
  2. Inert B-cell lymphoma (CLL, FL, MZL, LPL, HCL);
  3. Aggressive B-cell lymphoma (DLBCL, BL, MCL);
* Subject:

  1. Residual lesions remain after primary treatment and are not suitable for HSCT (Auto/Allo-HSCT);
  2. relapse after complete response (CR1) and unsuitable for allogeneic/autologous HSCT;
  3. Patients with high risk factors;
  4. relapse or no remission after hematopoietic stem cell transplantation or cellular immunotherapy.
* having measurable or evaluable lesions;
* The main tissues and organs of the patient function well:

  1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN);
  2. Renal function: creatinine < 220μmol/L;
  3. Lung function: indoor oxygen saturation ≥95%;
  4. Heart function: left ventricular ejection fraction (LVEF) ≥40%.
* Patients or their legal guardians voluntarily participate and sign the informed consent.

Exclusion Criteria:

* Pregnant or lactating women, or women who plan to become pregnant within six months;
* Infectious diseases (e.g. HIV, active hepatitis B or C infection, active tuberculosis, etc.);
* GVHD;
* Abnormal vital signs and failure to cooperate with the examination;
* People with mental or mental illness who are unable to cooperate with treatment and efficacy evaluation;
* People with high allergic constitution or severe allergic history, especially those allergic to IL-2;
* Subjects with systemic infection or severe local infection need anti-infection therapy;
* Complicated with dysfunction of heart, lung, brain, liver, kidney and other important organs;
* Any unstable systemic disease: including but not limited to unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥III);
* Doctors believe that there are other reasons for not being included in treatment.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Baseline up to 28 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
MRD negative overall response rate (MRD- ORR) | 3 months
  Assessment of MRD negative overall response rate (MRD- ORR) at 3 months of treatment
Overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 6, 12, 18 and 24
Event-free survival (EFS) | Month 6, 12, 18 and 24
  Assessment of EFS at Month 6, 12, 18 and 24
Overall survival (OS) | Month 6, 12, 18 and 24
  Assessment of OS at Month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, Ph.d, Study Chair — The Affiliated Hospital of Xuzhou Medical University; Junnian Zheng, Ph.D, Study Director — Xuzhou Medical University
Locations (1):
- The Affiliated hospital of Xuzhou medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No